CLINICAL TRIAL: NCT01253434
Title: E2022 Patch Formulation Single Dose Phase I Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2022-J081-001
Record Dates: First submitted 2010-11-30; First posted 2010-12-03 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2011-08

CONDITIONS: Japanese Healthy Male Adult Volunteers
Keywords: Transdermal Administration

ARMS (5):
- 1 (Experimental)
  Interventions: Drug: E2022
- 2 (Experimental)
  Interventions: Drug: E2022
- 3 (Experimental)
  Interventions: Drug: E2022
- 4 (Experimental)
  Interventions: Drug: E2022
- 5 (Experimental)
  Interventions: Drug: E2022

INTERVENTIONS:
Drug: E2022 — E2022 Type A patch
  Arms: 1
Drug: E2022 — E2022 Type B patch
  Arms: 2
Drug: E2022 — E2022 Type C patch
  Arms: 3
Drug: E2022 — E2022 Type D patch
  Arms: 4
Drug: E2022 — E2022 Type E patch
  Arms: 5

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of a single dose of E2022 in healthy Japanese male volunteers.

DETAILED DESCRIPTION:
This study is an open-label single site, randomized single dose study in 80 healthy Japanese male volunteers. The study consists of Period I to Period III, a total of 3 periods. In Period I, E2022 patches will be secured with seal. In Period II, single dose of E2022 5 mg tablet will be administered. In Period III, E2022 patches will be applied without seal. The features of the 5 patches will be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria

1. Body Mass Index (BMI) at Screening is 18.5 kg/m2 or above and less than 25.0 kg/m2: BMI (kg/m2)= weight(kg) ÷ {height(m)× height(m)}
2. Subjects who are between 20 and 55 years of age at the time of obtaining written consent.
3. Subjects who are willing to and can comply with the conditions described in the study protocol.

Exclusion Criteria

1. Subjects who consumed caffeine-containing food or beverages within 72 hours before study drug administration.
2. Exposure to any supplements or herbs (including Chinese medicine), or beverages (e.g. alcohol or grapefruit-containing beverages) known to modulate CYP3A4, CYP2C9, CYP2C19, CYP2D6, within 2 weeks before study drug administration.
3. Subjects with history of cutaneous hypersensitivity to external preparation, or those who are on another transdermal formulation.
4. Subjects who have excessive skin hair around the region to put the patch on.
5. Subjects with skin disorder, such as eczema, skin irritation, pigment disorder, injury or scar in the region of patch application, which may have an impact on skin findings.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Comparison of pharmacokinetics of E2022 patch (type A, B, C, D, E) with single dose of E2020 5 mg tablets. | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Tomoo Ogawa, Study Director — Neuroscience Clinical Development Section. JAC PCU. Eisai Co., Ltd.
Locations (1):
- Kagoshima, Kagoshima-ken, Japan